CLINICAL TRIAL: NCT00650663
Title: A Multicenter, Double-Blind, Randomized Study to Evaluate the Lipid-Altering Efficacy, Safety, and Tolerability of Ezetimibe Coadministered With Simvastatin Versus Simvastatin Monotherapy in African-American Subjects With Primary Hypercholesterolemia
Brief Title: Ezetimibe Plus Simvastatin Versus Simvastatin Alone in African-American Subjects With Primary Hypercholesterolemia (P03377)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P03377
Record Dates: First submitted 2008-03-31; First posted 2008-04-02 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia; Atherosclerosis
MeSH Terms: conditions — Hypercholesterolemia; Atherosclerosis | interventions — Ezetimibe, Simvastatin Drug Combination; Ezetimibe; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ezetimibe + Simvastatin (Experimental)
  Interventions: Drug: Ezetimibe + Simvastatin
- Simvastatin (Active Comparator)
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Ezetimibe + Simvastatin — oral tablets; ezetimibe 10 mg and simvastatin 20 mg once daily for 12 weeks
  Other Names: SCH 58235
  Arms: Ezetimibe + Simvastatin
Drug: Simvastatin — oral tablet; simvastatin 20 mg once daily for 12 weeks
  Arms: Simvastatin

SUMMARY:
The purpose of this study is to evaluate whether coadministration of ezetimibe 10 mg/day with simvastatin 20 mg/day for 12 weeks will result in greater reduction of LDL-C, total cholesterol (TC), triglycerides (TG), non HDL-C, and apolipoprotein B (ApoB), and greater increase in HDL-C, compared with simvastatin 20 mg/day as monotherapy for 12 weeks in African-American subjects with primary hypercholesterolemia. This study is being performed to better define the efficacy of ezetimibe coadministered with simvastatin in this population.

ELIGIBILITY:
Inclusion Criteria:

* Adult African-American or Black subjects with diagnosis of primary hypercholesterolemia with plasma LDL-C >=145 mg/dL and <=250 mg/dL, and plasma TG <=350 mg/dL
* Postmenopausal women who are receiving postmenopausal hormonal therapy or raloxifene must be maintained on a stable HRT or raloxifene regimen for at least 6 weeks and throughout the study
* Female subjects of non-childbearing potential
* Willingness to give written consent, participate and complete all study-related procedures, and ability to follow a stable NCEP Step I (or stricter) diet regimen and keep a diet diary when required.
* Clinical laboratory tests (CBC, blood chemistries, and urinalysis) within normal limits (except as noted below) or clinically acceptable.
* ALT (SGPT) and AST (SGOT) concentrations <=2 times the upper limit of normal (ULN) and creatine phosphokinase <=2 times the ULN.

Exclusion Criteria:

* Pregnancy or any other situation, condition, or illness that, in the opinion of the investigator, may interfere with optimal participation in the study
* Secondary forms of hyperlipidemia or underlying disease likely to limit life span to less than one year
* Known hypersensitivity or any contraindication to simvastatin or ezetimibe
* Use of investigational drugs within 30 days of study entry
* Concomitant illnesses: congestive heart failure NYHA Class III or IV; obstructive cardiomyopathy; uncontrolled cardiac arrhythmias; severe aortic stenosis; MI, CABG or angioplasty within 3 months of study; unstable or severe peripheral artery disease; unstable angina pectoris; study-limiting disorders of the hematologic, digestive or central nervous systems including cerebrovascular disease and degenerative disease; uncontrolled or newly diagnosed diabetes mellitus; uncontrolled endocrine or metabolic disease known to influence serum lipids or lipoproteins (clinically euthyroid subjects on stable replacement doses of thyroid hormone are eligible for enrollment); uncontrolled hypertension; known impairment of renal function (plasma creatinine >2.0 mg/dL), dysproteinemia, nephrotic syndrome or other renal disease (24-hour urinary protein 3+ or 1 gram); hepatobiliary or hepatic disease (AST or ALT >2 times the upper limit of the reference range); HIV positive; known coagulopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2003-10-01 (Actual); Primary Completion 2004-09-01 (Actual); Study Completion 2004-09-01 (Actual)

PRIMARY OUTCOMES:
Percent change in LDL-C from baseline to endpoint. | Week 12

SECONDARY OUTCOMES:
Percent change from baseline to endpoint in TC, TG, HDL-C, non-HDL-C, and ApoB. | Week 12

REFERENCES:
- [Result] Rodney RA, Sugimoto D, Wagman B, Zieve F, Kerzner B, Strony J, Yang B, Suresh R, Veltri E. Efficacy and safety of coadministration of ezetimibe and simvastatin in African-American patients with primary hypercholesterolemia. J Natl Med Assoc. 2006 May;98(5):772-8. PMID 16749654